CLINICAL TRIAL: NCT04909359
Title: Immunophenotypic Characterization of Crohn's Disease (CD) Responders to Vedolizumab
Brief Title: Characterization of CD Responders to Vedolizumab
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Maria Abreu, Professor of Medicine, University of Miami
Other Study IDs: 20150750; VEDO-IISR-2014-100892 (Other: Takeda)
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Crohn Disease; Ulcerative Colitis
Keywords: Inflammatory Bowel Disease (IBD); IBD; CD; UC; Vedolizumab; VDZ; Biomarkers; Response
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn's disease (CD): People with CD recently receiving vedolizumab as standard of care will be followed up to 5 years.
- Ulcerative colitis (UC): People with UC recently receiving vedolizumab as standard of care will be followed up to 5 years.

SUMMARY:
The purpose of this study is to characterize which patients with Crohn's disease are likely to respond to standard of care to vedolizumab therapy.

ELIGIBILITY:
Inclusion criteria:

1. Male or Female ≥18 and ≤70 years old.
2. Patients must be appropriate for baseline colonoscopy prior to induction therapy with vedolizumab.
3. Patients must have active inflammatory disease as seen by colonoscopy. 3A-Adult patients with moderately to severely active UC who have:

   1. had an inadequate response with, lost response to, or were;
   2. intolerant to a tumor necrosis factor (TNF) blocker or;
   3. immunomodulator; or had an inadequate response with, were;
   4. intolerant to, or demonstrated dependence on corticosteroids:

      * inducing and maintaining clinical response
      * inducing and maintaining clinical remission
      * improving endoscopic appearance of the mucosa
      * achieving corticosteroid-free remission 3B-Adult patients with moderately to severely active CD who have

   <!-- -->

   1. had an inadequate response with, lost response to, or were
   2. intolerant to a TNF blocker or immunomodulator; or had an
   3. inadequate response with, were intolerant to, or demonstrated
   4. dependence on corticosteroids:

      * achieving clinical response
      * achieving clinical remission
      * achieving corticosteroid-free remission
4. Patients will also have biochemical analysis with CRP and fecal calprotectin prior to initiating treatment with vedolizumab.

Exclusion criteria:

1. Patients that will not undergo colonoscopy at baseline prior to treatment with vedolizumab.
2. Patients who do not have endoscopic or biochemical (CRP, calprotectin) evidence of inflammation.
3. Patients that have been on natalizumab within 12 weeks of beginning vedolizumab.
4. Previous treatment with cyclosporine, thalidomide, or investigational drugs within 30 days of enrollment, prior treatment with vedolizumab
5. Toxic megacolon
6. Abdominal abscess
7. Symptomatic colonic stricture
8. Stoma
9. Increased risk of infection (eg, active or latent tuberculosis, immunodeficiency) Other clinically meaningful laboratory abnormalities: pregnancy or lactation, an unstable or uncontrolled medical disorder, colonic dysplasia or adenomas, and malignant neoplasms.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants being seen at the University of Miami IBD clinics with a diagnosis of CD or UC and about to initiate standard of care treatment with vedolizumab.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
T cell concentration | up to 22 weeks
  Evaluated from peripheral blood samples and lamina propria biopsies

SECONDARY OUTCOMES:
Effector memory T cells concentration | up to 22 weeks
  Evaluated from peripheral blood samples and lamina propria biopsies
T regulatory cells concentration | up to 22 weeks
  Evaluated from peripheral blood samples and lamina propria biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Abreu, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No